CLINICAL TRIAL: NCT02376621
Title: Nutrition Products - An Open-Label, Randomised, Single-Dose Study to Evaluate the Bioavailability of Omega-3 Based Dietary Supplements Under Fasting Conditions in Healthy Male and Female Subjects
Brief Title: Bioavailability of Omega-3 Food Supplements in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pronova BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: CTN00714102
Record Dates: First submitted 2015-02-11; First posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Healthy
Keywords: omega-3 based dietary supplements; Bioavailability
MeSH Terms: interventions — Triglycerides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- PronovaPure 150:500 triglycerides (Active Comparator): 3 × PronovaPure 150:500 triglycerides (TG) European Union (EU)
  Interventions: Dietary Supplement: PronovaPure 150:500 triglycerides; Dietary Supplement: Pronovum PRF-048; Dietary Supplement: Pronovum PRF-037; Dietary Supplement: PronovaPure 500:200 TG; Dietary Supplement: Pronovum PRF-047
- Pronovum PRF-048 (Active Comparator): 3 × Pronovum PRF-048
  Interventions: Dietary Supplement: PronovaPure 150:500 triglycerides; Dietary Supplement: Pronovum PRF-048; Dietary Supplement: Pronovum PRF-037; Dietary Supplement: PronovaPure 500:200 TG; Dietary Supplement: Pronovum PRF-047
- Pronovum PRF-037 (Active Comparator): 3 × Pronovum PRF-037
  Interventions: Dietary Supplement: PronovaPure 150:500 triglycerides; Dietary Supplement: Pronovum PRF-048; Dietary Supplement: Pronovum PRF-037; Dietary Supplement: PronovaPure 500:200 TG; Dietary Supplement: Pronovum PRF-047
- PronovaPure 500:200 TG (Active Comparator): 3 × PronovaPure 500:200 TG EU
  Interventions: Dietary Supplement: PronovaPure 150:500 triglycerides; Dietary Supplement: Pronovum PRF-048; Dietary Supplement: Pronovum PRF-037; Dietary Supplement: PronovaPure 500:200 TG; Dietary Supplement: Pronovum PRF-047
- Pronovum PRF-047 (Active Comparator): 3 × Pronovum PRF-047
  Interventions: Dietary Supplement: PronovaPure 150:500 triglycerides; Dietary Supplement: Pronovum PRF-048; Dietary Supplement: Pronovum PRF-037; Dietary Supplement: PronovaPure 500:200 TG; Dietary Supplement: Pronovum PRF-047

INTERVENTIONS:
Dietary Supplement: PronovaPure 150:500 triglycerides — Subjects will receive 5 single doses with at least 4 treatment-free days between each treatment period. The order of treatments will be in accordance with the randomisation schedule. Using a Williams design, 2 subjects will be randomly assigned to receive 1 of the following 10 treatment sequences:ABECD,BCADE, CDBEA, DECAB, EADBC, DCEBA, EDACB, AEBDC, BACED, CBDAE
Dietary Supplement: Pronovum PRF-048 — Subjects will receive 5 single doses with at least 4 treatment-free days between each treatment period. The order of treatments will be in accordance with the randomisation schedule. Using a Williams design, 2 subjects will be randomly assigned to receive 1 of the following 10 treatment sequences:ABECD,BCADE, CDBEA, DECAB, EADBC, DCEBA, EDACB, AEBDC, BACED, CBDAE
Dietary Supplement: Pronovum PRF-037 — Subjects will receive 5 single doses with at least 4 treatment-free days between each treatment period. The order of treatments will be in accordance with the randomisation schedule. Using a Williams design, 2 subjects will be randomly assigned to receive 1 of the following 10 treatment sequences:ABECD,BCADE, CDBEA, DECAB, EADBC, DCEBA, EDACB, AEBDC, BACED, CBDAE
Dietary Supplement: PronovaPure 500:200 TG — Subjects will receive 5 single doses with at least 4 treatment-free days between each treatment period. The order of treatments will be in accordance with the randomisation schedule. Using a Williams design, 2 subjects will be randomly assigned to receive 1 of the following 10 treatment sequences:ABECD,BCADE, CDBEA, DECAB, EADBC, DCEBA, EDACB, AEBDC, BACED, CBDAE
Dietary Supplement: Pronovum PRF-047 — Subjects will receive 5 single doses with at least 4 treatment-free days between each treatment period. The order of treatments will be in accordance with the randomisation schedule. Using a Williams design, 2 subjects will be randomly assigned to receive 1 of the following 10 treatment sequences:ABECD,BCADE, CDBEA, DECAB, EADBC, DCEBA, EDACB, AEBDC, BACED, CBDAE

SUMMARY:
The study will evaluate the bioavailability of omega-3 based dietary supplements under fasted conditions in healthy adult subjects. Each subject will participate in 5 treatment periods. The order of treatments will be in accordance with the randomisation schedule.There will be a minimum of 4 treatment-free days between each treatment period. On each dosing occasion, subjects will be fasted for at least 10 hours overnight, prior to the morning of dosing. Twenty-four subjects will be enrolled to complete dosing of 20 subjects.

ELIGIBILITY:
Inclusion Criteria:

* males or females
* any ethnic origin
* age 40 - 65 years
* BMI 18.5 - 30.0 kg/m2
* generally in good health
* signed informed consent

Exclusion Criteria:

* males or females not willing to use appropriate contraception
* prescribed systemic or topical medication taken within 14 days
* taken supplements containing omega-3 faty acids or fish oil last 14 days or any non-prescribed systemic or topical medication including herbal remedies and vitamin/mineral supplements within 7 days
* taken any medication including St. John's Worth known to alter drug absorption within 30 days
* subjects participating in a clinical study past 3 months
* recent blood donation
* significant history of drug allergy or any allergic disease
* allergy or hypersensitivity to omega-3 fatty acids, fish, soya, oleic acid, sesame oil or other constituents of pharmaceutical preparation.
* high consumption of tobacco
* high consumption of alcohol
* other significant medical history or physical findings (including HIV,hepatitis)
* vegetarians
* not willing to follow dietary restrictions
* frequent migraine attacks
* previously taken part in or withdrawn from study or according to investigator should not participate.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Area under curve of omega-3 based dietary supplements under fasted conditions. | Pharmacokinetics up to 36 hours postdose
Peak plasma concentration of omega-3 based dietary supplements under fasted conditions. | Pharmacokinetics up to 36 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Brooks, MD, Principal Investigator — Covance Clinical Research Unit (CRU) Ltd.
Locations (1):
- Covance Clinical research Unit (CRU) Ltd,Springfield House, Hyde street, Leeds, United Kingdom